CLINICAL TRIAL: NCT03104595
Title: EC-18 for Management of Chemotherapy-Induced Neutropenia in Patients With Advanced BC Receiving Low Febrile Neutropenia Risk Chemotherapy: Dose-Escalation, Open-label, Trial to Assess Safety and Tolerability of EC-18
Brief Title: Management of Severe Chemotherapy-induced Neutropenia in Advanced Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Enzychem Lifesciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EC-18-201
Record Dates: First submitted 2017-02-24; First posted 2017-04-07 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Febrile Neutropenia
Keywords: EC-18, febrile neutropenia, breast cancer, chemotherapy
MeSH Terms: conditions — Febrile Neutropenia; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 3 + 3 dose escalation
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): EC-18 500 mg
  Interventions: Drug: EC-18
- Cohort 2 (Experimental): EC-18 1000 mg
  Interventions: Drug: EC-18
- Cohort 3 (Experimental): EC-18 1500 mg
  Interventions: Drug: EC-18
- Cohort 4 (Experimental): EC-18 2000 mg
  Interventions: Drug: EC-18
- Cohort 5 (Experimental): EC-18 3000 mg
  Interventions: Drug: EC-18
- Cohort 6 (Experimental): EC-18 4000 mg
  Interventions: Drug: EC-18

INTERVENTIONS:
Drug: EC-18 — oral administration
  Other Names: EC-18 soft capsules

SUMMARY:
To assess the safety and establish the dose to assess the pharmacokinetic activity following administration of EC-18 in patients with advanced breast cancer receiving low febrile neutropenia risk chemotherapy who are the candidates for second-line or higher combination therapy with doxorubicin and cyclophosphamide.

DETAILED DESCRIPTION:
This study will utilize a non-randomized, open-label 3 + 3 dose escalation design in which subjects will receive 500 mg, 1000 mg, 1500 mg, 2000 mg, 3000 mg and 4000mg of EC-18. The stepwise daily dosing by cohort was performed for 21 days (3 weeks)

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥19 years of age
2. Subjects who have voluntarily signed the informed consent prior to the screening tests to participate in the study
3. Subjects who have been diagnosed as adenocarcinoma of the breast and relapsed after adjuvant or primary (neoadjuvant) chemotherapy, and was confirmed based on documented medical history to be candidates for second-line or higher combination chemotherapy with doxorubicin and cyclophosphamide to treat relapsed or metastatic disease.
4. Subjects with adequate function of major organs based on the following clinical laboratory values in the latest test performed within 28 days prior to IP dosing:

   * Neutrophil count (ANC): ≥1,500/mm3
   * Platelet count: ≥10.0×10^4/mm3
   * Hemoglobin: ≥9.0 g/dL
   * AST, ALT: ≤3.0 x ULN
   * Serum total bilirubin: ≤1.5 mg/dL
   * Serum creatinine: ≤1.5 mg/dL
5. Subjects whose Eastern Cooperative Oncology Group (ECOG) performance score is 0-1.
6. For women of child bearing potential, subjects should have willingness to use acceptable contraceptive methods during the entire clinical study period.
7. Subjects who are capable of understanding the overall procedure of the clinical study and are willing to participate in compliance with all test procedures.

Exclusion Criteria:

1. Subjects with active and inactive hepatitis, patients with history of HIV, or other uncontrolled infectious disease.
2. Subjects with a history of HIV positive or currently undergoing/received antiretroviral therapy, and subjects with a history of hepatitis B surface antigen positive, or current positive hepatitis C disease.
3. Subjects who received radiation therapy within 4 weeks prior to assignment to treatment group.
4. Subjects who have been diagnosed within 5 years with other types of cancer except for those who have been appropriately treated for superficial non-melanoma skin cancer or cervical intraepithelial neoplasia.
5. Subjects with a history of intolerance for granulocyte colony stimulating factor treatment
6. Subjects who are expected to show hypersensitivity to the IP or its ingredients
7. Subjects with a positive urine pregnancy test result at screening visit or before the first administration of the study drug
8. Subjects who took any other investigational product in other clinical study within 30 days prior to screening visit.
9. Clinically significant unstable medical abnormality; psychiatric disorder, chronic disease, alcohol or drug use disorder, or other significant biological, psychological, or social factor, which in the investigator's opinion, unfavorably affects the risk-benefit ratio of study participation or likely to affect study results.
10. Subjects with heart disease (i.e. congestive heart failure, arrhythmia, symptomatic coronary artery disease); Myocardial infarction within 6 months before initiation of the study.
11. Subjects with left ventricular ejection fraction (LVEF) < 50% at screening.
12. Significant neurological or psychiatric disorders including dementia or seizures.
13. Patients with dyslipidemia not controlled by drugs [based on LDL-C and TG levels for which treatment is recommended by the Korean dyslipidemia treatment guidelines and the U.S. National Cholesterol Education Program-Adult Treatment Panel III]
14. Uncontrolled diabetes mellitus (HbA1c >7%; if the level is confirmed after 6 months or longer treatment with oral hypoglycemic agents or insulin)
15. Subjects who have received systemic chemotherapy with doxorubicin to treat metastatic or recurrent breast cancer
16. Subjects with grade 2 or higher peripheral sensory neuropathy at screening visit or before the first dosing of the study drug
17. Subjects who have undergone significant gastrectomy along with intractable nausea and vomiting, chronic gastrointestinal disease, or clinically significant sequelae, which would interfere with proper absorption of the study drug
18. Subjects who administered systemic antibiotics within 14 days prior to administration of the study drug
19. Subjects whose cumulative dose of doxorubicin exceeded 240 mg/m2
20. Subjects who were currently receiving trastuzumab

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 28 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Duration of Grade 4 neutropenia | 15 days after starting chemotherapy
  Complete blood count and absolute neutrophil count assessed daily to determine febrile neutropenia

SECONDARY OUTCOMES:
Incidence of Grade 3-4 neutropenia | For 15 days after starting chemotherapy (except Day 3 and 4)
  The grade for Neutropenia is assessed according to NCI CTCAE 4.03 version
Incidence of febrile neutropenia | For 15 days after starting chemotherapy (except Day 3 and 4)
  Febrile neutropenia is assessed by ANC and body temperature according to NCI CTCAE version 4.03

OTHER OUTCOMES:
Incidence of adverse events | 3-week treatment period and follow-up visit at day 36
  Incidence of treatment-emergent adverse events, serious adverse events, adverse events leading to discontinuation, adverse events by severity grade
Clinical laboratory evaluations | 3-week treatment period and follow-up visit at day 36
  Clinical laboratory tests (hematology, clinical chemistry, coagulation, and urine test result analysis) -- absolute values and changes from the baseline
Vital signs | 3-week treatment period and follow-up visit at day 36
  Absolute values and changes from baseline in vital signs
12-lead electrocardiogram (ECG) | 3-week treatment period and follow-up visit at day 36
  Absolute values and changes from baseline ECG

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Bae Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - National Cancer Center, Gyeonggi-do
  - Yonsei University Health System Severance Hospital, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No